CLINICAL TRIAL: NCT03622827
Title: Postoperative Concurrent Chemoradiotherapy Combined With Recombinant Human Endostatin for High-risk Early Stage Cervical Cancer: A Phase II Pilot Study (ChESS).
Brief Title: Postoperative Concurrent Chemoradiotherapy Combined With Endostar for High-risk Early Stage Cervical Cancer
Acronym: ChESS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing Medical University (Other)
Collaborators: Second Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, Ke Gu, Associate professor, Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K2018009
Record Dates: First submitted 2018-07-31; First posted 2018-08-09 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Uterine Cervical Neoplasms
Keywords: Adjuvant therapy; chemoradiotherapy; Uterine Cervical Neoplasms; high risk; Endostar
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chemoradiotherapy + Endostar (Experimental): Chemoradiotherapy with Endostar：
  * Chemoradiotherapy: pelvic radiotherapy with concurrent chemotherapy that consisted of cisplatin (75 mg/m2, day 1-3) and 5-fluorouracil (5-FU; 1000mg/m2/day,civ, day 1-4) for 2 cycles every 3 weeks.
  * Endostar: recombinant human endostatin (15mg/m2/d, civ, d1-7) is given 3 days before the chemotherapy every 3 weeks, total of two cycles during chemoradiotherapy course.
  Interventions: Combination Product: Chemoradiotherapy+ Endostar

INTERVENTIONS:
Combination Product: Chemoradiotherapy+ Endostar — Chemoradiotherapy with Endostar：
  * Chemoradiotherapy: pelvic radiotherapy starts 2-3 weeks after surgery. Intensity modulated radiotherapy (IMRT) is given five fractions per week at 1.8-2 Gy/fraction/day with total dose summed up to 45-50Gy. The external beam radiotherapy should be completed within 6 weeks.
  * Concurrent chemotherapy is consisted of cisplatin (75 mg/m2, day 1-3) and 5-fluorouracil (5-FU; 1000mg/m2/day, civ, day 1-4) for 2 cycles every 3 weeks.
  * Endostar: recombinant human endostatin (15mg/m2/d, civ, d1-7) is given 3 days before the concurrent chemoradiotherapy for 2 cycles every 3 weeks.

SUMMARY:
To assess the efficacy and safety of postoperative concurrent chemoradiotherapy combined with recombinant human endostatin (Endostar) in patients with high-risk early stage cervical cancer.

DETAILED DESCRIPTION:
This is a pilot phase 2, single arm study to assess the efficacy and safety of concurrent chemoradiotherapy combined with recombinant human endostatin (Endostar) in early stage cervical cancer patients with high risk factor(s).

Postoperative pelvic radiotherapy starts 2-3 weeks after surgery. Intensity modulated radiotherapy (IMRT) is given five fractions per week at 1.8-2 Gy/fraction/day with total prescription dose of 45-50Gy to PTV region. The external beam radiotherapy should be completed within 6 weeks. Concurrent chemotherapy consists of cisplatin (75 mg/m2, day 1-3) and 5-fluorouracil (5-FU; 1000mg/m2/day, civ, day 1-4) for 2 cycles every 3 weeks. Recombinant human endostatin (Endostar,15mg/m2/d, civ, d1-7) is applied 3 days before the concurrent chemoradiotherapy for 2 cycles every 3 weeks.

Aimed to recruit total of 120 cases in this single arm study. The primary endpoint is 3-year disease-free survival and acute toxicity. Secondary endpoints include time to distant metastasis survival, local-regional recurrence free survival, 3 and 5-year overall survival, and safety and tolerability. Quality of life will be evaluated with EORTC-Q30.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 70 years.
* Histologically confirmed adenocarcinoma or squamous cervical carcinomas.
* Chest CT scan and ultrasound must be done prior to surgery as to rule out distant metastasis.
* Operable patients with clinical diagnosis of FIGO stage IB-IIA cervical cancer.
* Complete radical hysterectomy of cervical cancer is mandatory. All gross diseases must have been removed at the end of surgery. All surgical margins of resection must be negative for tumor. Para-aortic lymph node sampling is performed according to gynaecologist decision.
* Patients with one of these risk factors:positive pelvic nodes, parametrial invasion, positive surgical margin.OR patients with at least two of following risk factors: tumor size≥4cm,lymphovascular space invasion,stromal invasion≥1/2.
* Performance status 0-2 (ECOG, Eastern Cooperative Oncology Group).
* Adequate organ function is needed, including cardio-respiratory, hepato-renal and hematological reserves: Absolute neutrophil count (ANC)≥1.5×109/L;Platelet count≥100×109/L; ASAT&ALST<1.5 times upper limit of normal (ULN) (With hepatic metastases, ASAT&ALST<5.0 times upper limit of normal);Bilirubin <1.5 times ULN;Creatinine≤1.25×ULN or Creatinine clearance≥50 mL/min.
* Signed written informed consent prior to study entry.

Exclusion Criteria:

* Previous radiation or chemotherapy treatment or major pelvic surgery.
* Patients with distant metastasis confirmed by imaging or pathology.
* Other uncured malignant tumors in the past five years, except the cured skin basal cell carcinoma and breast carcinoma in situ.
* Any prior anticancer therapy.
* Unable to tolerate postoperative concurrent chemoradiotherapy.
* Patients with evidence of being allergic to fluorouracil, cisplatin or Endostar.
* Patients with serious comorbidity that might potentially influence the practice of protocol, including severe infection, myocardial infarction, severe arrhythmia, severe cerebrovascular disease, severe mental disorder, etc.
* Patients with Heart related adverse events or thrombotic events in the past 6 months.
* Patients with hepatitis B, hepatitis C and human immunodeficiency virus (HIV) or any other active viral infections.
* Participate in other clinical researchers.
* The estimated survival<3 months;

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-07-31 (Actual); Primary Completion 2023-07-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
3-year Disease-free survival | 3 years
  From date of surgery until the date of first documented local-regional progression or distant metastasis (determined by CT or MRI scan and/or biopsy) or death (from any cause) assessed up to three years.
Acute toxicity | 3 months
  Evaluate the treatment induced toxicity according to CTCAE 4.0 during the time of chemoradiotherapy and Endostar which starts from the first day of Endostar and lasts three months.

SECONDARY OUTCOMES:
Time to distant metastasis survival | 3 years
  Determine the non-distant metastasis survival in early-stage cervical cancer patients with high risk factors, defined as time from the date of surgery to first distant metastasis event (determined by CT or MRI scan and/or pathologic disease on biopsy).
Local-regional recurrence free survival | 3 years
  Determine the local-regional recurrence free survival in early-stage cervical cancer patients with high risk factors, defined as time from the date of surgery to first local-regional recurrence event (determined by CT or MRI scan and/or pathologic disease on biopsy).
3-year overall survival rate | 3 years
  Determine the 3-year overall survival rate in early-stage cervical cancer patients with high risk factors, defined as time from the date of surgery to death of all cause at time of 3 years after operation.
5-year overall survival rate | 5 years
  Determine the 5-year overall survival rate in early-stage cervical cancer patients with high risk factors, defined as time from the date of surgery to death of all cause at time of 5 years after operation.
Quality of Life (QoL) | 3 years
  Collect QoL data on early-stage cervical cancer patients with high risk factors. The data is measured by EORTC QLQ-C30 (Version 3.0) according to investigator collection at the starting and ending time of the adjuvant treatment. EORTC QLQ-C30 is a questionnaire developed to assess the quality of life of cancer patients. The core and disease-specific for cervix modules are selected to estimate treatment related influence on patients' life. The final score of the questionnaire is collected and analyzed according to detailed scoring procedures from manuals.

CONTACTS AND LOCATIONS:
Overall Officials: Ke Gu, M.D., Ph.D, Principal Investigator — The Affiliated Suzhou Hospital of Nanjing Medical University
Locations (1):
- The Affiliated Suzhou Hospital of Nanjing Medical University, Suzhou, Jiangsu, China